CLINICAL TRIAL: NCT05658367
Title: Effect of Massage Made With Aromatherapy Oil After Mastectomy on Acute Arm Pain and Anxiety: a Randomized Controlled Study
Brief Title: Effect of Aromatherapy Massage on Pain and Anxiety After Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: mataseven
Record Dates: First submitted 2022-12-02; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-03

CONDITIONS: Acute Pain; Anxiety; Mastectomy; Massage Therapy; Aromatherapy
MeSH Terms: conditions — Acute Pain; Anxiety Disorders | interventions — Sesame Oil; Massage

STUDY DESIGN:
Intervention Model Description: The research was carried out to determine the effect of aromatherapy arm massage with sesame oil, sesame-lavender oil mixture, and paraffin oil on acute pain severity and anxiety level in women who underwent Interventional Simple Mastectomy (BM)/Modified Radical Mastectomy (MRM). The study design arm is three groups and a randomized controlled, double-blind, drug-free clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Although there is information in the literature that it is not possible to blind the participants due to the characteristic smell of aromatherapy oils, patients are shown blind in aromatherapy massage because the oils are formulated and the oil content is not known by the patients (Nasiri and Farsi, 2017; Rasooli et al., 2016). Due to the feasibility and nature of the study, the principal investigator cannot be blinded during grouping, while blinding will be provided for the patients and the analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): - Group I: The group applied arm massage with sesame oil
  Interventions: Procedure: Aromatherapy massage with sesame oil
- Group 2 (Experimental): - Group II: The group applied arm massage with a mixture of sesame-lavender oil
  Interventions: Procedure: Aromatherapy massage with sesame- lavender oil mixed
- Group 3 (Placebo Comparator): - Group III (Control): The group applied arm massage with paraffin oil
  Interventions: Procedure: Massage with parraffin oil

INTERVENTIONS:
Procedure: Aromatherapy massage with sesame- lavender oil mixed — After the surgery, 3 hours after the painkiller application, the patients will massage their arms with sesame- lavender oil mixed for 15 minutes with classical massage manipulations.
  Other Names: Group 1
  Arms: Group 2
Procedure: Aromatherapy massage with sesame oil — After the surgery, 3 hours after the painkiller application, the patients will massage their arms with sesame oil for 15 minutes with classical massage manipulations.
  Other Names: Group 2
  Arms: Group 1
Procedure: Massage with parraffin oil — After the surgery, 3 hours after the painkiller application, the patients will massage their arms with paraffin oil for 15 minutes with classical massage manipulations.
  Other Names: Group 3 (Placebo- Control)
  Arms: Group 3

SUMMARY:
This study is an interventional type three-group randomized controlled non-drug clinical trial aimed at targeting the acute pain content and anxiety level of aromatherapy arm treatment with a sesame oil and sesame lavender oil mixture performed with Simple Mastectomy (BM) / Modified Radical Mastectomy (MRM). It constitutes a total of 66 patients with the power to represent the universe. However, considering the losses that may occur during the study process, it was decided that it would be appropriate to include 90 patients, 36% more than the sample. Individuals receiving arm massage with sesame oil (Group I), individuals performing arm massage with sesame-lavender oil mixture (Group II), and individuals performing arm massage with paraffin oil (Group III) constitute the research groups. After obtaining the informed written consent of the participants who agreed to participate in the study, the randomization list created from the computer-based random numbers table will be used with the block randomization method to assign an equal number of people to all three groups. In the preoperative period, patients will be given an allergic sensitivity (patch) test of the oils to be used in the study to Groups 1 and 2, massage training will be given to all groups with the show-and-have method in the pre-operative period, a massage application brochure and video will be given, and information will be given on how to fill out the follow-up forms. H1: After Simple Mastectomy (BM)/Modified Radical Mastectomy (MRM), massage with sesame oil reduces the severity of acute arm pain compared to massage with paraffin oil.H2: After simple mastectomy (BM)/Modified Radical Mastectomy (MRM), massage with a sesame-lavender oil mixture reduces the severity of acute arm pain compared to massage with paraffin oil.H3: After Simple Mastectomy (BM)/Modified Radical Mastectomy (MRM), massage with sesame oil reduces anxiety levels compared to massage with paraffin oil.H4: After Simple Mastectomy (BM)/Modified Radical Mastectomy (MRM), massage with a sesame-lavender oil mixture reduces anxiety levels compared to massage with paraffin oil.H5: After Simple Mastectomy (BM)/Modified Radical Mastectomy (MRM), massage with a sesame-lavender oil mixture reduces the severity of acute arm pain compared to massage with sesame oil.H6: After Simple Mastectomy (BM)/Modified Radical Mastectomy (MRM), massage with a sesame-lavender oil mixture reduces anxiety levels compared to massage with sesame oil.

DETAILED DESCRIPTION:
Breast cancer ranks first among the most common cancers in women in Turkey, and one out of every four women diagnosed in 2014 was breast cancer (Turkish Ministry of Health Public Health Institution, Turkey Cancer Statistics, 2017). Breast cancer is considered both a local and systemic disease. In the planning of the treatment, the decision of surgery is made by considering the stage of cancer, and the most frequently applied intervention is mastectomy, which involves the partial or complete removal of the breast tissue (Turkish Ministry of Health, General Directorate of Health Services. Breast Cancer Prevention, Screening, Diagnosis, Treatment, and Follow-up Clinical Guide, 2020; Tola et al., 2021). It is stated that in patients who have undergone breast surgery, especially during axillary lymph node dissection, due to the possibility of intercostobrachial nerve injury, pain, numbness, and weakness may be felt in the chest wall, arm, and shoulder in the postoperative period, acute/chronic, neuropathic and phantom pain, lymphedema may develop (Ozmen, 2012; Nemli et al., 2017). Post-operative pain decreases in the first few days, but in some patients, the severity of pain does not decrease or even increase despite post-operative pain management (Mc Mahon et al., 2013). Anxiety experienced by patients in the preoperative period, including breast cancer patients, is an important factor in the level of pain intensity felt after surgery (Stamenkovic et al., 2018; Kulkarni et al., 2017). Effective anxiety and acute pain management are important in terms of shortening the recovery period of the individual, reducing the treatment costs, preventing the occurrence of chronic pain, and increasing the quality of life. For this reason, it is mentioned that non-pharmacological methods can be used in addition to pharmacological treatment to assist treatment (Chou et al., 2016; Small and Laycock, 2020; Reisli et al., 2021). Today, it is known that aromatherapy has an important place among complementary and holistic therapy methods (Zor et al., 2021). However, it is stated that the studies on aromatherapy massage are weak in terms of evidence and more studies should be done on this subject (Ayik and Ozden, 2018). It is stated that aromatherapy oils are applied by inhalation method alone rather than applied with massage, there are few studies on the effectiveness of massage with aromatic oils, therefore more studies on aromatherapy massage should be done in the treatment of pain, anxiety, and depression (Crosby, 2018; Raffi, 2020).

It is seen that studies conducted after breast surgery are mostly focused on the development of chronic pain rather than acute pain intensity after surgery (Kulkarni et al., 2017). In the literature, the effects of aromatherapy massage on anxiety and acute pain severity in patients who are planning for breast surgery are examined, foot reflexology or classical massage (Dion et al., 2015) according to the massage area preferred by the patient in the postoperative period, classical massage applied to the chest region in the preoperative period (Dion et al., 2015). Xiao et al., 2018) there is research on interventions.

No clinical study was found that evaluated the severity of acute pain and anxiety level in the arm after Simple Mastectomy (SM) / Modified Radical Mastectomy (MRM) surgery with sesame oil, sesame-lavender oil mixture, and aromatherapy massage applied in the postoperative period. Therefore, the result of this study is important because it forms the basis for a clinical study.

With the results to be obtained from the research; It is aimed at better understanding the effects of these herbal-based agents in aromatherapy treatment, contributing to nurses' non-pharmacological treatment interventions, and providing quality care in the management of anxiety and acute pain in patients, and thus to provide new information to evidence-based nursing practices.

ELIGIBILITY:
Inclusion criteria;

* 18 years and over,
* literate,
* Agreeing to participate in the study,
* Person, place, and time orientation,
* Visual (except for those with better vision using a visual aid), auditory communication difficulties (except for those with better hearing ability using a hearing aid) that will prevent them from understanding the information given and expressing the pain situation correctly,
* No speech impediment/communication problem,
* Simple mastectomy (BM) and modified radical mastectomy (MRM) were performed,
* Not using any TAT method,
* Able to use technology (smartphone, computer, etc.),
* Individuals with technology devices (smartphone, tablet, computer, etc.)

Exclusion criteria;

* Not speaking Turkish and illiterate in Turkish,
* Those who are allergic to the oils to be used in the massage during the application,
* Involved in a different study conducted in the clinic,
* Breast prosthesis placed during surgery,
* Having physical and cognitive problems at a level that cannot apply massage,
* Individuals diagnosed with mood disorders (using any medication for depression, panic attacks, dysthymia, or bipolar disorder)
* Transferred to the intensive care unit in the postoperative period,
* Severe bleeding, hematoma, seroma, nerve injury, or lymphedema developing in the postoperative period,
* Developing an allergy to the oils to be used in the massage during the application,
* Those who want to leave work voluntarily,
* Individuals who do not comply with the working process and conditions will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is the most frequently diagnosed type of cancer among women worldwide, and breast cancer ranks first among the most common cancers in women.
Enrollment: 90 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Change in NUMERICAL PAIN SCALE (NUMERİCAL RATING SCALE- NRS) | In the postoperative period, the patient's pain is recorded at 08:00 and 08:30, 20:00 and 20:30 with analgesic application, and at 11:00, 11:15 and 23:00 and 23:15 with massage application.
  It is based on the expression of pain intensity in numbers. In numerical scales, 0 points define the absence of pain, while the value of the number increases as the severity of pain increases, and 10 points indicate unbearable pain
STATUS ANXIETY SCALE | Instant anxiety data of the patient are recorded in the postoperative period, at the 15th minute after the massage.
  It is a 20-item scale used to measure the instantaneous anxiety level of individuals.

SECONDARY OUTCOMES:
VITAL FINDINGS REGISTRATION FORM | In the postoperative period, the patient's body temperature is recorded 0 minutes before the analgesic, 30 minutes after the analgesic, 0 minutes before the massage and 15 minutes after the massage.
  It is the form that includes the patient's body temperature.
ANALGESIC FOLLOW-UP FORM | Data are taken from the patient's file during the hospitalization for 2 days.
  In this form, information about the name, type, number/dose, route of administration and frequency of analgesic administered in the postoperative period is included.
VITAL FINDINGS REGISTRATION FORM | In the postoperative period, the patient's pulse is recorded 0 minutes before the analgesic, 30 minutes after the analgesic, 0 minutes before the massage and 15 minutes after the massage.
  It is the form that includes the patient's pulse.
VITAL FINDINGS REGISTRATION FORM | In the postoperative period, the patient's respiratory is recorded 0 minutes before the analgesic, 30 minutes after the analgesic, 0 minutes before the massage and 15 minutes after the massage.
  It is the form that includes the patient's respiratory.
VITAL FINDINGS REGISTRATION FORM | In the postoperative period, the patient's blood pressure is recorded 0 minutes before the analgesic, 30 minutes after the analgesic, 0 minutes before the massage and 15 minutes after the massage.
  It is the form that includes the patient's blood pressure.

OTHER OUTCOMES:
NUMERICAL PAIN SCALE (NUMERİCAL RATING SCALE- NRS) | The patient's pain is recorded in the preoperative period.
  It is based on the expression of pain intensity in numbers. In numerical scales, 0 points define the absence of pain, while the value of the number increases as the severity of pain increases, and 10 points indicate unbearable pain
STATUS ANXIETY SCALE | Instant anxiety data of the patient are recorded in the preoperative period.
  It is a 20-item scale used to measure the instantaneous anxiety level of individuals.
VITAL FINDINGS REGISTRATION FORM | The body temperature of the patient are recorded in the preoperative period.
  It is the form that includes the patient's body temperature.
VITAL FINDINGS REGISTRATION FORM | The pulse of the patient are recorded in the preoperative period.
  It is the form that includes the patient's pulse.
VITAL FINDINGS REGISTRATION FORM | The respiratory of the patient are recorded in the preoperative period.
  It is the form that includes the patient's respiratory.
VITAL FINDINGS REGISTRATION FORM | The blood pressure of the patient are recorded in the preoperative period.
  It is the form that includes the patient's blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Muzeyyen Ataseven, Principal Investigator — Istanbul Marmara Universty; Nuray Sahin Orak, Study Director — Istanbul Nisantasi University
Locations (2):
- Turkey (Türkiye) (2):
  - Sisli Etfal Training and Research Hospital, Istanbul, Eyalet/Yerleşke
  - Sisli Etfal Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No